CLINICAL TRIAL: NCT00901706
Title: Multidimensional Assessment and Intervention for Elder Self-Neglect
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: The Center for Clinical and Translational Sciences (CCTS) Clinical Research Unit at The University of Texas Health Science Center at Houston (Other)
Responsible Party: Principal Investigator, Carmel Dyer, Professor, Internal Medicine, Geriatrics, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HSC-MS-08-0052
Record Dates: First submitted 2009-05-12; First posted 2009-05-14 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Self-Neglect; Cognitive Ability, General; Geriatric Disorder
Keywords: Self-Neglect; Comprehensive Geriatric Assessment (CGA); Geriatric Syndromes; Quality of Life; Basic Activities of Daily Living; Instrumental Activities of Daily Living
MeSH Terms: interventions — Geriatric Assessment; Randomized Controlled Trials as Topic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CGA plus APS Usual Care (Experimental): Comprehensive geriatric assessment coupled with Adult Protective Services (APS) usual care for elders with self-neglect.
  Interventions: Other: Comprehensive Geriatric Assessment and APS Usual Care; Other: APS usual care
- APS Usual Care (Active Comparator): APS usual care consisting of social, medical, and legal interventions.
  Interventions: Other: Comprehensive Geriatric Assessment and APS Usual Care; Other: APS usual care

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment and APS Usual Care — Comprehensive Geriatric Assessment coupled with APS usual care which collectively will consist standardized cognitive, functional, affective, social, and legal interventions.
  Other Names: Randomized Controlled Trial
Other: APS usual care — APS usual care consists of social, medical, and legal assistance.
  Other Names: Randomized Controlled Trial

SUMMARY:
This study is designed to assess the best method for caring for elders reported to Adult Protective Services (APS) for self-neglect. Specifically, this study will compare APS usual care coupled with interdisciplinary comprehensive geriatric care to APS usual care alone in improving the health and quality of live among elders with substantiated self-neglect.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* English Speaking
* Resident of Harris County, Houston Texas
* Community-dwelling
* Substantiated Self-Neglect

Exclusion Criteria:

* No other substantiated allegations
* Non-community dweller
* No available for projected follow-up period
* Impaired decision-making with no available proxy
* Already receiving care from TEAM or within the past year
* Terminal Illness

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-08; Primary Completion 2012-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Self-Neglect Severity Scale (SSS) | Baseline and 6-months

SECONDARY OUTCOMES:
Functional Status | Baseline and 6-months
Kohlman Evaluation of Living Skills (KELS) | Baseline and 6-months
Mini-mental State Exam (MMSE) | Baseline and 6-months
15-item Geriatric Depression Scale | Baseline and 6-months
Physical Performance Test (PPT) | Baseline and 6-months
SF-36 Health Survey | Baseline and 6-months
The Duke Social Support Index (DSSI) | Baseline and 6-months
Client Satisfaction Questionnaire (CSQ-8) | Baseline and 6-months
Costs of Social Services and Health Care Utilization and Costs | Months 1,2,3,4,5,6

CONTACTS AND LOCATIONS:
Overall Officials: Carmel B. Dyer, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States